CLINICAL TRIAL: NCT06809569
Title: A Pilot Study to Evaluate the Use of Laser Speckle Contrast Imaging on Changes in Dermal Blood Flow Induced by Intradermal Capsaicin and Topical AITC in Healthy Participants
Brief Title: A Study to Evaluate Laser Speckle Contrast Imaging to Assess Changes in Chemical Agent-Induced Skin Blood Flow in Healthy Participants (MK-0000-420)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0000-420; MK-0000-420 (Other: MSD)
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — allyl isothiocyanate; Capsaicin; 2,3,4-tri-O-acetylarabinopyranosyl isothiocyanate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laser Speckle Contrast Imaging (Experimental): Participants receive topical Allyl Isothiocyanate (AITC) application and intradermal capsaicin application sequentially along with a placebo comparator (vehicle for AITC and vehicle for capsaicin) once every 2 weeks per protocol to perform laser speckle contrast imaging.
  Interventions: Drug: Allyl Isothiocyanate (AITC); Drug: Capsaicin; Other: Vehicle for AITC; Other: Vehicle for Capsaicin

INTERVENTIONS:
Drug: Allyl Isothiocyanate (AITC) — Topical administration
Drug: Capsaicin — Intradermal administration
Other: Vehicle for AITC — Topical administration
Other: Vehicle for Capsaicin — Intradermal administration

SUMMARY:
Pain is a significant issue and there is a need for better treatments for pain management. Local changes in skin blood flow can be used as an indicator of pain in the body. Capsaicin and allyl isothiocyanate (AITC) increase blood flow and cause pain. The purpose of this study is to evaluate the use of laser speckle contrast imaging (LSCI) as a tool to assess changes in skin blood flow. Researchers want to learn about the effect size and reproducibility of using LSCI to measure the blood flow response to capsaicin and AITC.

ELIGIBILITY:
Inclusion Criteria:

* Is in good health based on medical history, physical examination, vital sign measurements, and electrocardiograms performed before randomization
* Has a skin surface without significant skin allergies, pigmentary disorders or active dermatological conditions that may interfere with the conduct of the laser speckle contrast imaging (LSCI) assessment

Exclusion Criteria:

* Has a history of clinically significant endocrine, gastrointestinal, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases
* Has a history of stroke, chronic seizures, epilepsy, peripheral neuropathy or other clinically significant neurological disease or cognitive impairment that are severe enough to interfere with assessment of pain (sensory) systems

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Mean Dermal Blood Flow (DBF) in the Region of Interest (ROI) | Up to approximately 60 minutes
  DBF is defined as the local changes in the skin blood flow after application of study intervention. DBF will be measured via a Laser Speckle Contrast Imager. The mean DBF in the ROI will be reported.
Area Under the Curve from Time 0 to 20 Minutes (AUC0-20) of Mean DBF in the ROI | Up to approximately 20 minutes
  AUC0-20 is defined as the area under the curve from time 0-20 minutes. DBF is defined as the local changes in the skin blood flow after application of study intervention. DBF will be measured via a Laser Speckle Contrast Imager. AUC0-20 of mean DBF in ROI will be reported.
Area Under the Curve from Time 0 to 60 Minutes (AUC0-60) of Mean DBF in the ROI | Up to approximately 60 minutes
  AUC0-60 is defined as the area under the curve from time 0-60 minutes. DBF is defined as the local changes in the skin blood flow after application of study intervention. DBF will be measured via a Laser Speckle Contrast Imager. AUC0-60 of mean DBF in ROI will be reported.

SECONDARY OUTCOMES:
Change from Baseline in the Mean Intensity of DBF (Flare-1 Mean) | Baseline, Up to 60 minutes
  Flare-1 mean is defined as the mean perfusion of measurement points exceeding baseline mean DBF + 1 standard deviation. The change from baseline in the mean intensity of DBF (Flare-1 Mean) will be reported.
Change from Baseline in the Area of DBF (Flare-1 Area) | Baseline, Up to 60 minutes
  Flare-1 area is defined as the total area of points with perfusion values exceeding baseline mean DBF + 1 standard deviation. The change from baseline in the area of DBF (Flare-1 Area) will be reported.
Change from Baseline in the Mean Intensity of DBF (Flare-2 Mean) | Baseline, Up to 60 minutes
  Flare-2 mean is defined as the mean perfusion of points with perfusion values exceeding baseline mean DBF + 2 standard deviations. The change from baseline in the mean intensity of DBF (Flare-2 Mean) will be reported.
Change from Baseline in the Area of DBF (Flare-2 Area) | Baseline, Up to 60 minutes
  Flare-2 area is defined as total area of points with perfusion values exceeding baseline mean DBF + 2 standard deviations. The change from baseline in the area of DBF (Flare-2 Area) will be reported.
Mean Change From Baseline in Pain Intensity Measured Using a Pain Numeric Rating Scale (NRS) | Baseline, Up to 60 minutes
  The participant's pain intensity will be assessed on each arm utilizing a pain numeric rating scale (NRS). NRS will characterize pain on a scale of 0 to 10, with 0 being 'no pain' and 10 being the 'worst pain' imaginable. The higher score indicates worse pain intensity. The mean change from baseline in pain intensity will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Center for Clinical Pharmacology (CCP) (Site 0001), Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com